CLINICAL TRIAL: NCT06943768
Title: Fecal DNA Methylation and Helicobacter Pylori Gastric Cancer Susceptibility Genes for the Early Diagnosis and Screening of Gastric Cancer
Brief Title: Fecal DNA Methylation and Helicobacter Pylori Gastric Cancer Susceptibility Genes Test
Status: Not yet recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Dazhi Xu, Director of the gastric surgery department, Fudan University
Other Study IDs: 2410-Exp092
Record Dates: First submitted 2025-03-20; First posted 2025-04-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2024-11

CONDITIONS: Gastric (Stomach) Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: fecal methylation site-based testing and fecal Helicobacter pylori gastric cancer susceptibility gene-based testing — To establish an early diagnostic test system for gastric cancer based on the methylation site detection technology in feces, with or without the combination of Helicobacter pylori gastric cancer susceptibility gene detection, and then to evaluate the clinical diagnostic value of this test system.

SUMMARY:
This is a multicenter, cross-sectional study. It is based on fecal methylation site detection, H. pylori susceptibility testing of fecal samples, and a combination of the two, compared with the "gold standard" imaging tests, CT, gastroscopy and/or pathology, for gastric cancer, benign diseases such as gastritis, and health check-ups.

DETAILED DESCRIPTION:
Primary study objective: to evaluate the sensitivity and specificity of fecal methylation site-based and fecal Helicobacter pylori gastric cancer susceptibility gene assays applied to early diagnosis and screening of gastric cancer.

Secondary research objectives: 1. the accuracy, kappa value, area under the ROC curve, positive likelihood ratio, negative likelihood ratio, positive predictive value, and negative predictive value of fecal methylation site-based testing and fecal Helicobacter pylori gastric cancer susceptibility gene-based testing applied for predicting gastric cancer; 2. whether the predictive ability is significantly higher than that of conventional tumor markers, such as CA19-9, CEA, and CA72-4; and 3. the follow up of Gastritis and healthy people, to assess the cases of gastric cancer during the follow-up period and the clinical diagnosis and treatment prediction; 4. Follow-up gastric cancer patients, to assess the association with gastric cancer recurrence metastasis and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old, male or female not limited.
* Within 90 days, the gastroscopy and/or pathological results confirm the absence of gastric cancer.
* Patients must be able to fully understand the informed consent form and be able to personally sign it.

Exclusion Criteria:

* Severe cardiac, hepatic, or renal insufficiency, or psychiatric disorders.
* A previous history of malignant tumors of the upper gastrointestinal tract.
* Women during pregnancy.
* Those with undefined pathology.
* Those with unsatisfactory sample retention (e.g., too small a sample size)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The subjects of this clinical study are from the community population in the high incidence area of gastric cancer in Tongling. The subjects will collect feces during medical visits or physical examinations, and undergo fecal methylation DNA and Helicobacter pylori gastric cancer susceptibility gene testing. The researchers determine the study subjects based on the inclusion and exclusion criteria and inform them of the content of the informed consent form.
Sampling Method: Probability Sample
Enrollment: 9654 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity | Baseline
  Sensitivity and specificity of fecal DNA methylation detection and Helicobacter pylori gastric cancer susceptibility genes based on their application for early diagnosis and screening of gastric cancer.